CLINICAL TRIAL: NCT06103786
Title: Effects of High-Intensity Interval Training on Physical Fitness, Skills, and Tactical Performance Among College Male Ice Hockey Players In China
Brief Title: Effects of High-Intensity Interval Training on Physical Fitness, Skills, and Tactical Performance, 12 Weeks High-Intensity Interval Training
Acronym: HIIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Yuan Yandong, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Yuan Yandong
Record Dates: First submitted 2023-08-07; First posted 2023-10-27 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Power, Personal
Keywords: High-intensity interval training; Physical fitness; Skills; Tactical performance

STUDY DESIGN:
Intervention Model Description: This experiment utilized a high-intensity interval training methodology to intervene in the physical fitness, skills, and tactical performance of college athletes and compared it to traditional technical skill training methods.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Repeated Sprint 2. Interval Sprint 3.Long-Pass Tracking Drill 4. Chase-The-Rabbit Tracking Drill (Experimental): 1. Make repeated sprints on the ice for a certain distance to measure its speed.
  2. On the ice, perform 15 seconds of intermittent acceleration on the ice, with 30 seconds between each slide.
  3. On the ice, make a long pass before taking a shot, then turn to track back.
  4. On the ice, skate down the ice, 2 on 1, with a puck to pass and shoot.
  Interventions: Behavioral: Assigned Interventions
- 1. Varied Pace Skating 2.Driblling and Shooting Drill 3. Passing and Catching training 4. 2-on-1 (Experimental): 1. On the ice, a 1-minute accelerated skate and skating at an even pace for 2 minutes
  2. On the ice, dribbling the ball and shooting at the goal
  3. On the ice, they stood facing each other at a distance of 20 meters and practiced passing and catching.
  4. On the ice, practice 2-on-1 offensive tactics and complete shots on goal.
  Interventions: Behavioral: Random Interventions

INTERVENTIONS:
Behavioral: Assigned Interventions — Ice hockey players did 12 weeks of on-ice high-intensity interval training. Their training included:
  Repetitive sprint training Sprint interval training Long-pass tracking drills Chase-the-rabbit tracking drills High-intensity interval training in four types improved college ice hockey players' sports performance in 12 weeks.
  Arms: 1. Repeated Sprint 2. Interval Sprint 3.Long-Pass Tracking Drill 4. Chase-The-Rabbit Tracking Drill
Behavioral: Random Interventions — Ice hockey players did 12 weeks of traditional on-ice training. Their training included:
  Varied pacing skating Dribbling and shooting Passing and catching drills 2-on-1 offensive tactics Traditional training in four types improved college ice hockey players' sports performance in 12 weeks.
  A 12-week on-ice training program was conducted on college players to observe its effects on their physical fitness, skills, and tactical performance compared to an experimental and control group.
  Arms: 1. Varied Pace Skating 2.Driblling and Shooting Drill 3. Passing and Catching training 4. 2-on-1

SUMMARY:
This clinical trial aims to compare the difference between high-intensity interval training and common traditional training on physical fitness, skills, and tactical performance among college ice hockey players in China.

The main questions it aims to answer are:

* 1. How does high-intensity interval training affect the physical fitness of college ice hockey players?
* 2. How does high-intensity interval training affect the skills of college ice hockey players?
* 3. How does high-intensity interval training affect the tactical performance of college ice hockey players? Participants will be asked to do 12 weeks of high-intensity interval training and common traditional training to see if there are differences between the two and the positive effects of high-intensity interval training.

DETAILED DESCRIPTION:
Through experimental design and quantitative research methods. This experiment will test the effectiveness of the training method by intervening in the selective fitness, skills, and tactical performance of college students using a high-intensity interval training method on the ice. The experiment will use 12 weeks of high-intensity interval training to improve the fitness, skills, and tactical performance of the intervention for ice hockey players. The experiment consists of two groups, with 20 students in the experimental group and 20 students in the control group, to compare the differences between the two groups. The experiment was divided into a discussion group and a general teaching group. The purpose of this experiment is to provide a theoretical basis for the improvement of ice hockey training methods so that college ice hockey players can obtain better competitive performance, especially in physical fitness and technique.

The experimental group (1-12 weeks) performed repeated sprint training, sprint interval training (on-ice 45-s shift length conditioning drill), a long-pass tracking drill, and a chase-the-rabbit tracking drill. There are three phases: 1-4 weeks, 5-8 weeks, and 9-12 weeks, gradually increasing the intensity of training. Similarly, the control group performed varied-pace skating (1 minute accelerated skating, 2 minutes even pace), dribbling and shooting drill (30 m), passing-catching drill (20 m), and 2 on 1 offensive drill (full rink). As in the experimental group, the same three phases were used to gradually increase the intensity.

ELIGIBILITY:
Inclusion Criteria:

1. College male ice hockey players aged from 18 to 24.
2. Athletes from HPU and AXU universities: the experimental group in the training base of Henan Polytechnic University, and the control group in the training base of Anhui Xinhua.

Exclusion Criteria:

1. Recent (less than 1 year) history of knee, elbow, waist, or shoulder injury: History of rheumatic disease or nerve injury and still receiving treatment.
2. Participate in high-intensity interval training before the study.
3. According to the requirements of the coach, participants with light motivation, negative training attitude and no willingness to participate in repeated training and testing were selected during the completion of the experimental task.
4. Athletes directly interrupt training due to some factors.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2023-11-20 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake performance among collegiate ice hockey players | before the experiment
  1. Maximum oxygen uptake measured during intensity training at 90-95% of maximum heart rate (per minute, per kilogram of body weight, the maximum amount of oxygen obtained (milliliters) will be combined to report VO2 max in ml/kg-min), #ml/kg-min#
The endurance performance of college ice hockey players | before the experiment
  1. The endurance level of the athletes was assessed using the Yo-Yo Intermittent Recovery Test Level 1 scale. The evaluation range is 5-23 points; the higher the score, the higher the endurance level.
The power performance of college ice hockey players | before the experiment
  1. A countermovement jump and a squat jump evaluate the power. The higher the jump, the stronger the power, #cm#
The agility and skill performance of college ice hockey players | before the experiment
  1. Using the Illinois Agility Test method of assessing athlete agility, the shorter the time, the higher the agility, #s#
  2. The time to skate to 20- and 30-meter, #s#
  3. The time to skate 20 meters with the ball, #s#
The passing and shooting performance of college ice hockey players | before the experiment
  1. Number of passes at distance 20m each other in a minute, #pcs#
  2. Number of successful shots on goal in one minute, #pcs#
Tactical performance among college ice hockey | before the experiment
  1. Evaluate the effect of attacking tactics by the number of shots and goals scored. The more shots and goals scored, the better the tactical effect.
  2. The offensive tactics were assessed based on the level of cooperation among players, their proficiency, and their success rate in passing and receiving. The coordination fluency was evaluated using a scale ranging from 1 to 10, where higher scores indicated greater fluency. The success rate was determined by calculating the percentage of successful passes out of the total passes made, multiplied by 100. Higher values reflected a higher success rate.

SECONDARY OUTCOMES:
Maximum oxygen uptake performance of college ice hockey players | 6 weeks end
  1. Maximum oxygen uptake measured during intensity training at 90-95% of maximum heart rate (per minute, per kilogram of body weight, the maximum amount of oxygen obtained (milliliters) will be combined to report VO2 max in ml/kg-min), #ml/kg-min#
The endurance performance of college ice hockey players | 6 weeks end
  1. The endurance level of the athletes was assessed using the Yo-Yo Intermittent Recovery Test Level 1 scale. The evaluation range is 5-23 points; the higher the score, the higher the endurance level.
The power performance of college ice hockey players | 6 weeks end
  1. A countermovement jump and a squat jump evaluate the power. The higher the jump, the stronger the power, #cm#
The agility and skill performance of college ice hockey players | 6 weeks end
  1. Using the Illinois Agility Test method of assessing athlete agility, the shorter the time, the higher the agility, #s#
  2. The time to skate to 20- and 30-meter, #s#
  3. The time to skate 20 meters with the ball, #s#
The passing and shooting performance of college ice hockey players | 6 weeks end
  1. Number of passes at distance 20m each other in a minute, #pcs#
  2. Number of successful shots on goal in one minute, #pcs#
Tactical performance among college ice hockey | 6 weeks end
  1. Evaluate the effect of attacking tactics by the number of shots and goals scored. The more shots and goals scored, the better the tactical effect.
  2. The offensive tactics were assessed based on the level of cooperation among players, their proficiency, and their success rate in passing and receiving. The coordination fluency was evaluated using a scale ranging from 1 to 10, where higher scores indicated greater fluency. The success rate was determined by calculating the percentage of successful passes out of the total passes made, multiplied by 100. Higher values reflected a higher success rate.

OTHER OUTCOMES:
Maximum oxygen uptake performance of college ice hockey players | 12 weeks end
  1. Maximum oxygen uptake measured during intensity training at 90-95% of maximum heart rate (per minute, per kilogram of body weight, the maximum amount of oxygen obtained (milliliters) will be combined to report VO2 max in ml/kg-min), #ml/kg-min#
The endurance performance of college ice hockey players | 12 weeks end
  1. The endurance level of the athletes was assessed using the Yo-Yo Intermittent Recovery Test Level 1 scale. The evaluation range is 5-23 points; the higher the score, the higher the endurance level.
The power performance of college ice hockey players | 12 weeks end
  1. A countermovement jump and a squat jump evaluate the power. The higher the jump, the stronger the power, #cm#
The agility and skill performance of college ice hockey players | 12 weeks end
  1. Using the Illinois Agility Test method of assessing athlete agility, the shorter the time, the higher the agility, #s#
  2. The time to skate to 20- and 30-meter, #s#
  3. The time to skate 20 meters with the ball, #s#
The passing and shooting performance of college ice hockey players | 12 weeks end
  1. Number of passes at distance 20m each other in a minute, #pcs#
  2. Number of successful shots on goal in one minute, #pcs#
Tactical performance among college ice hockey | 12 weeks end
  1. Evaluate the effect of attacking tactics by the number of shots and goals scored. The more shots and goals scored, the better the tactical effect.
  2. The offensive tactics were assessed based on the level of cooperation among players, their proficiency, and their success rate in passing and receiving. The coordination fluency was evaluated using a scale ranging from 1 to 10, where higher scores indicated greater fluency. The success rate was determined by calculating the percentage of successful passes out of the total passes made, multiplied by 100. Higher values reflected a higher success rate.

CONTACTS AND LOCATIONS:
Overall Officials: YANDONG YUAN, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Yuan Yandong, Jiaozuo, Henan, China

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate.

REFERENCES:
- [Background] Buchheit M, Laursen PB. High-intensity interval training, solutions to the programming puzzle. Part II: anaerobic energy, neuromuscular load and practical applications. Sports Med. 2013 Oct;43(10):927-54. doi: 10.1007/s40279-013-0066-5. PMID 23832851
- See also: This article is from National Library of Medinice — https://pubmed.ncbi.nlm.nih.gov/23832851/